CLINICAL TRIAL: NCT03584906
Title: Comparison of Graft Quality and Patient Morbidity Following Four Different Connective Tissue Graft Harvesting Techniques. A Randomized Controlled Feasibility Study
Brief Title: Comparison of Graft Quality and Patient Morbidity Following Palatal Harvesting.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Giulio Rasperini, Professor of Periodontology, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Palatal Harvesting and CTG
Record Dates: First submitted 2018-06-19; First posted 2018-07-12 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Gingival Recession; Palate; Wound
MeSH Terms: conditions — Gingival Recession; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- De-epithelialized gingival graft (DGG) (Experimental): A harvesting approach where the a graft is obtained from the superficial palate and then extra-orally de-epithelialized in order to obtain a connective tissue graft (DGG harvesting approach) Then the DGG is used for treating gingival recessions (root coverage procedure)
  Interventions: Procedure: DGG Harvesting approach; Procedure: Root coverage procedure
- Envelope technique (ET) (Experimental): A harvesting approach where only one horizontal incision is performed on the palate (ET harvesting approach) for harvesting a connective tissue graft.
  Then the connective tissue graft is used for treating gingival recessions (root coverage procedure)
  Interventions: Procedure: ET harvesting approach; Procedure: Root coverage procedure
- Trap door technique (TDT) (Experimental): A harvesting approach where one horizontal and two vertical incisions are performed on the palate (TDT harvesting approach) for harvesting a connective tissue graft.
  Then the connective tissue graft is used for treating gingival recessions (root coverage procedure)
  Interventions: Procedure: TDT harvesting approach; Procedure: Root coverage procedure
- Maxillary tuberosity (MT) (Experimental): A harvesting approach that obtains an epithelialized gingival graft from the maxillary tuberosity (MT harvesting approach) which is then extra-orally de-epithelialized in order to obtain a connective tissue graft.
  Then the connective tissue graft is used for treating gingival recessions (root coverage procedure)
  Interventions: Procedure: MT harvesting approach; Procedure: Root coverage procedure

INTERVENTIONS:
Procedure: DGG Harvesting approach — An epithelialized graft is harvested from the superficial palate and then extraorally de-epithelialized in order to obtain a connective tissue graft
  Arms: De-epithelialized gingival graft (DGG)
Procedure: ET harvesting approach — A connective tissue graft is harvested from the palate after reflecting a primary palatal flap
  Arms: Envelope technique (ET)
Procedure: TDT harvesting approach — A connective tissue graft is harvested from the palate after reflecting a primary palatal flap
  Arms: Trap door technique (TDT)
Procedure: MT harvesting approach — An epithelialized graft is harvested from the maxillary tuberosity and then extraorally de-epithelialized in order to obtain a connective tissue graft
  Arms: Maxillary tuberosity (MT)
Procedure: Root coverage procedure — A single or multiple gingival recession is treated with a coronally advanced flap and a connective tissue graft

SUMMARY:
The purpose of this study is to compare four different connective tissue graft harvesting technique in terms of graft quality and patient post-operative morbidity

DETAILED DESCRIPTION:
The primary aim is to compare 4 different connective tissue graft harvesting techniques in terms of morbidity and in terms of quality of the graft.

The secondary aim is to evaluate the outcome of gingival recessions treated with grafts obtained from different harvesting approaches, in terms of mean root coverage, complete root coverage, keratinized tissue gain, clinical attachment level gain and gingival thickness

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater,
* Patients with no reported systemic diseases,
* Healthy periodontium or demonstrating stable periodontal condition following conventional periodontal therapy,
* Full mouth plaque score (FMPS) and full mouth bleeding score (FMBS) of < 15%,
* Clinical indication for periodontal plastic surgery utilizing CTG to treat either a single or a maximum of two recession defects (Miller class I, II) around natural teeth
* No history of previous palatal harvesting

Exclusion Criteria:

* Pregnancy
* Systemic condition that generally precludes surgical therapy or that could influence the outcome of therapy (e.g. Diabetes with HbA1c > 7%, INR > 3 etc.)
* Non-compensated systemic disease
* Poor oral hygiene with full mouth plaque score (FMPS) and full mouth bleeding score (FMBS) > 20% at baseline
* Inadequate endodontic treatment or tooth mobility at the site of surgery
* Radiographic evidence of bone loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Patient morbidity (VAS) | 14 days
  Patient post-operative pain measured using a VAS scale
Mean root coverage (mRC) | 6 months
  mRC measured as a percentage

SECONDARY OUTCOMES:
Clinical attachment level (CAL) gain | 6 months
  CAL gain measured in mm
Gingival thickness (GT) | 6 months
  CAL gain measured in mm
Patient willingness for retreatment | 14 days
  Patient willingness for retreatment (related to graft harvesting), if necessary, expressed as "yes" or "no"
Painkillers consumption | 14 days
  Painkiller consumption expressed in mg
Root coverage Esthetic Score (RES) | 6 months
  RES measured using numeric values from 0 to 10
Keratinized tissue (KT) gain | 6 months
  KT gain measured in mm

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Rasperini, DDS, Principal Investigator — University of Milan
Locations (2):
- Italy (2):
  - University of Milan, Milan
  - Studio Odontoiatrico, Piacenza

REFERENCES:
- [Background] Zucchelli G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, de Sanctis M. Patient morbidity and root coverage outcome after subepithelial connective tissue and de-epithelialized grafts: a comparative randomized-controlled clinical trial. J Clin Periodontol. 2010 Aug 1;37(8):728-38. doi: 10.1111/j.1600-051X.2010.01550.x. Epub 2010 Jun 24. PMID 20590963
- [Background] Tavelli L, Barootchi S, Nguyen TVN, Tattan M, Ravida A, Wang HL. Efficacy of tunnel technique in the treatment of localized and multiple gingival recessions: A systematic review and meta-analysis. J Periodontol. 2018 Sep;89(9):1075-1090. doi: 10.1002/JPER.18-0066. Epub 2018 Aug 13. PMID 29761502
- [Background] Tavelli L, Ravida A, Saleh MHA, Maska B, Del Amo FS, Rasperini G, Wang HL. Pain perception following epithelialized gingival graft harvesting: a randomized clinical trial. Clin Oral Investig. 2019 Jan;23(1):459-468. doi: 10.1007/s00784-018-2455-5. Epub 2018 Apr 30. PMID 29713890
- [Background] Wessel JR, Tatakis DN. Patient outcomes following subepithelial connective tissue graft and free gingival graft procedures. J Periodontol. 2008 Mar;79(3):425-30. doi: 10.1902/jop.2008.070325. PMID 18315424
- [Background] Lorenzana ER, Allen EP. The single-incision palatal harvest technique: a strategy for esthetics and patient comfort. Int J Periodontics Restorative Dent. 2000 Jun;20(3):297-305. PMID 11203571